CLINICAL TRIAL: NCT01324895
Title: Retrospective Analysis of Treatment Outcomes in Patients With Bacterial Overgrowth Syndrome Diagnosed by D-Xylose Breath Testing
Acronym: SIBO
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 406-2010
Record Dates: First submitted 2011-03-24; First posted 2011-03-29 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Small Intestinal Bacterial Overgrowth Syndrome (SIBO); Small Bowel Bacterial Overgrowth Syndrome (SBBOS)
Keywords: Small intestinal bacterial overgrowth syndrome (SIBO); bacterial overgrowth syndrome; Small Bowel Bacterial Overgrowth Syndrome (SBBOS); 14-Co2 D-Xylose Breath Testing; Antibiotics; Prokinteics; Prokinetic Agents
MeSH Terms: conditions — Blind Loop Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to compare the efficacy of prokinetics versus antibiotics versus a combination of antibiotics plus prokinetics in the eradication of Small-Intestinal Bacterial Over-Growth Syndrome (SIBO) in those with and without a positive D-xylose Breath Test.

Hypothesis: Patients with SIBO treated with a combination of prokinetics and in particular octreotide and antibiotics will have reduced recurrence rates of SIBO than either therapy given alone.

DETAILED DESCRIPTION:
We want to determine whether treatment with prokinetics such as Octreotide, Azithromycin, Erythromycin or Tegaserod alone, versus antibiotics alone, or combination of antibiotics plus prokinetics results in symptomatic improvement in patients with SIBO (defined by a positive D xylose Breath test).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had 14 C-D-Xylose Breath test performed in GI Motility Laboratory at the University of Florida

Exclusion Criteria:

* Those who cannot tolerate 14 C-D-Xylose Breath test for any reason

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have had 14 C-D-Xylose Breath test performed in GI Motility Laboratory at the University of Florida to help define the cause of their symptoms and for diagnosis of SIBO, between January 2000 up until the date of IRB approval.
Sampling Method: Non-Probability Sample
Enrollment: 944 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
clinical response to treatments as measured by changes in patients' GI symptoms, weight and lab data | A retrospective chart review of up to 8 clinical visits between January 2000 and September 2010 will be conducted on all patients who have had a D-Xylose Breath Test at the Shands Motility Laboratory at the University of Florida during this time period
  Overall clinical response to each treatment (antibiotic, pro-kinetic, or both) and any symptoms reported in up to 8 separate clinical visits in the follow-up of these patients during the above mentioned time period will be analyzed and reviewed retrospectively using the patients' charts.

CONTACTS AND LOCATIONS:
Overall Officials: Baharak Moshiree, MD, MS, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Singh VV, Toskes PP. Small Bowel Bacterial Overgrowth: Presentation, Diagnosis, and Treatment. Curr Treat Options Gastroenterol. 2004 Feb;7(1):19-28. doi: 10.1007/s11938-004-0022-4. PMID 14723835
- [Background] Lombardo L, Foti M, Ruggia O, Chiecchio A. Increased incidence of small intestinal bacterial overgrowth during proton pump inhibitor therapy. Clin Gastroenterol Hepatol. 2010 Jun;8(6):504-8. doi: 10.1016/j.cgh.2009.12.022. Epub 2010 Jan 6. PMID 20060064
- [Background] King CE, Toskes PP, Spivey JC, Lorenz E, Welkos S. Detection of small intestine bacterial overgrowth by means of a 14C-D-xylose breath test. Gastroenterology. 1979 Jul;77(1):75-82. No abstract available. PMID 447030
- [Background] Pimentel M. Review of rifaximin as treatment for SIBO and IBS. Expert Opin Investig Drugs. 2009 Mar;18(3):349-58. doi: 10.1517/13543780902780175. PMID 19243285
- [Background] Attar A, Flourie B, Rambaud JC, Franchisseur C, Ruszniewski P, Bouhnik Y. Antibiotic efficacy in small intestinal bacterial overgrowth-related chronic diarrhea: a crossover, randomized trial. Gastroenterology. 1999 Oct;117(4):794-7. doi: 10.1016/s0016-5085(99)70336-7. PMID 10500060
- [Background] Verne GN, Eaker EY, Hardy E, Sninsky CA. Effect of octreotide and erythromycin on idiopathic and scleroderma-associated intestinal pseudoobstruction. Dig Dis Sci. 1995 Sep;40(9):1892-901. doi: 10.1007/BF02208652. PMID 7555439
- [Background] Soudah HC, Hasler WL, Owyang C. Effect of octreotide on intestinal motility and bacterial overgrowth in scleroderma. N Engl J Med. 1991 Nov 21;325(21):1461-7. doi: 10.1056/NEJM199111213252102. PMID 1944424
- [Background] Lauritano EC, Gabrielli M, Scarpellini E, Lupascu A, Novi M, Sottili S, Vitale G, Cesario V, Serricchio M, Cammarota G, Gasbarrini G, Gasbarrini A. Small intestinal bacterial overgrowth recurrence after antibiotic therapy. Am J Gastroenterol. 2008 Aug;103(8):2031-5. doi: 10.1111/j.1572-0241.2008.02030.x. PMID 18802998